CLINICAL TRIAL: NCT03528070
Title: A Clinical Study of Tranilast in the Treatment of Sarcoidosis
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FirstNanjingMUMH Hou
Record Dates: First submitted 2018-04-19; First posted 2018-05-17 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2018-01

CONDITIONS: Sarcoidosis
Keywords: Sarcoidosis; Tranilast; skin; lung
MeSH Terms: conditions — Sarcoidosis | interventions — tranilast

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tranilast (Experimental)
  Interventions: Drug: Tranilast

INTERVENTIONS:
Drug: Tranilast — Subjects will be treated with tranilast

SUMMARY:
56 patients with sarcoidosis will be selected to receive treatment of tranilast.The investigators can analyse the changes in the thickness and area of skin lesions before and after treatment as well as other involved organs nodule size changes to determine the efficacy and safety of drugs.

DETAILED DESCRIPTION:
56 patients with sarcoidosis will be selected. After the signing of the informed consent ,participants will be collected the initial lesions photos, the size of the lump by ultrasound, the forced vital capacity(FVC), and chemical examinations including blood routine examination, routine urine test, liver function, renal function. During tranilast treatment (0.1g each time, three times a day) , participants need regular follow-up (1 per month) including liver and kidney function, blood glucose level monitoring, every three months to retest ultrasound and the forced vital capacity(FVC). With 3 month as a time point, participants were observed for four points(one point if only skin invasion ).After the experiment, the experimental data will be arranged and the data will be statistically processed (t test) to determine whether it is meaningful.

ELIGIBILITY:
Inclusion Criteria:

* (1)patients with diagnosed sarcoidosis, the skin pathology showed non necrotic granuloma and negative staining of fungi and atypical mycobacterium; (2)No corticosteroids and immunosuppressants were used for nearly 1 months.

Exclusion Criteria:

* 1)with a liver or kidney disease, or accompanied by a tumor or a severe infection ; (2)with mental disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2018-05 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Changes in the size of the pulmonary nodule by ultrasound | 12 months
  During tranilast (0.1g each time, three times a day,12 months) treatment, patients need to retest the size of the pulmonary nodule by ultrasound. The investigators can get the changes in the size of the pulmonary nodule.
Changes of the forced vital capacity(FVC) | 12 months
  During tranilast (0.1g each time, three times a day,12 months) treatment, patients need to retest the forced vital capacity(FVC),then get the changes.